CLINICAL TRIAL: NCT02581540
Title: Mersey Acute Coronary Syndrome Rule-Out Using High Sensitive Troponin (MACROS) : A Comparison of Risk Scores in Consecutive, Unselected Chest Pain Presentations With Suspected Acute Coronary Syndrome in the Era of High Sensitive Troponin
Brief Title: Mersey Acute Coronary Syndrome Rule-Out Using High Sensitive Troponin
Acronym: MACROS
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 808/15
Record Dates: First submitted 2015-07-20; First posted 2015-10-21 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2016-08

CONDITIONS: Acute Coronary Syndrome; Angina Pectoris; Cardiovascular Diseases; Chest Pain; Heart Diseases; Myocardial Ischemia; Heart Attack; Chest Pain Atypical Syndrome; Angina, Unstable; Myocardial Infarction
Keywords: Troponin; High Sensitivity Troponin T; MACE; risk stratification; suspected cardiac chest pain; Acute Coronary Syndrome; GRACE; TIMI; HEART
MeSH Terms: conditions — Acute Coronary Syndrome; Angina Pectoris; Cardiovascular Diseases; Chest Pain; Heart Diseases; Myocardial Ischemia; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected Cardiac Chest Pain: This cohort is observed for the incidence of MACE (death, non-fatal myocardial infarction and emergency revascularisation)

SUMMARY:
The aim of this observational study is twofold. The primary hypothesis being tested is that initial(first) high sensitivity Tn <5ng/l (limit of detection) combined with an ECG with no ischaemic changes is superior as an accelerated diagnostic tool/strategy compared to TIMI score (<2), GRACE <75 and HEART score ≤ 3. (Hs tn T- Roche elecsys HS tn T) and also against HS troponin at the 99th percentile (<15ng/l with nonischaemic changes)- again all scored with initial (first tn ) only.

The second aim is to directly compare the three established methods of risk stratifying patients (predicting risk in suspected heart attacks) namely, the Global Registry of Acute Coronary Events (GRACE), Thrombolysis in Myocardial Infarction (TIMI) and HEART score in the era of high sensitivity troponins performs best.

DETAILED DESCRIPTION:
Chest pain results in up to 9.4% of presentations to emergency departments in the UK and up to 27.4% of hospital admissions. The morbidity, mortality and economic costs associated with this constitute a significant burden on the National Health Service (NHS). Distinguishing patients with serious and potentially life-threatening causes of chest pain from those with 'benign' causes is important but often difficult.

There are numerous risk stratification scores available for estimating risk in patients with heart attacks but these have not been widely applied or tested in those presenting to accident and emergency department with chest pain when the diagnosis of a heart attack has not yet been established but is suspected. These tools were based on conventional Troponin assays. The advent of the new Elecsys highly-sensitive (HS) Troponin T assays has led to improved and earlier detection of heart attacks. high sensitivity refers to analytic sensitivity - much lower concentrations of troponin can be identified in the blood.

The aim of this prospective observational cohort study is twofold. Firstly to determine whether the results of a single high sensitivity troponin and electrocardiogram (ECG) could be used alone to direct care (expedite early discharge in those ECG and troponin negative). A discharge strategy of high sensitive troponin (<5ng/l) with a nonsichaemic ECG will be directly compared to the following: hs troponin at or below the 99th percentile (<15ng/l) + a nonischaemic ECG, TIMI score <2, HEART score ≤ 3 and GRACE score <75.

Secondly we wish to determine which of the three established methods of risk stratifying patients (predicting risk in suspected heart attacks) namely, the Global Registry of Acute Coronary Events (GRACE), Thrombolysis in Myocardial Infarction (TIMI) and HEART score in the era of HS troponin T performs best.

Patients presenting to the emergency department at Aintree University Hospital, Merseyside between June 2011 and October 2011 with suspected cardiac chest pain are prospectively recruited and information entered into an electronic database. The study comprises of 1750 consecutive patients (3056 with chest pain but only 1750 with suspected cardiac chest pain). All data collated will form the basis for risk stratification scores (GRACE, TIMI, HEART) calculation. These risk scores will give a predicted event rate (death, heart attack, stenting procedure or bypass).

The main outcome measures are major adverse cardiac events(MACE)- death, non-fatal myocardial infarction and emergency revascularisation at 6 weeks, and 1 year. the outcomes will be blinded (to initial risk scores) and independently adjudicated by consultant cardiologists with a 3rd consultant cardiologist experienced in clinical endpoint adjudication used to resolve differences.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged >18 years presenting to the emergency department at Aintree University Hospital,Merseyside between June-November 2011 with suspected cardiac chest pain

Exclusion Criteria:

* The presence of a definitive non-ischaemic cause for chest pain, trauma-related chest pain, cardiac arrest on arrival to the ED.
* Patients without HS troponin T which indicates no suspicion of a cardiac cause of chest pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department at a single large teaching hospital- Aintree University Hospital, Merseyside between June 2011 and November 2011 with suspected cardiac chest pain
Sampling Method: Probability Sample
Enrollment: 3054 (Actual)
Dates: Start 2011-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with major adverse cardiac events(MACE)- death, non-fatal myocardial infarction and emergency revascularisation at 1 year | 12 months observational period from recruitment date
  To compare the observed versus predicted incidence of major adverse cardiovascular events (MACE) amongst the three methods of risk stratifications (GRACE, TIMI, HEART) at 1 year in order to determine the most effective risk score

SECONDARY OUTCOMES:
Number of Participants with major adverse cardiac events(MACE)- death, non-fatal myocardial infarction and emergency revascularisation ; in patients with a normal ECG/initial Troponin | 12 months observational period from recruitment date
  To determine if the combination of a negative high sensitivity troponin T and a normal ECG at presentation is associated with a lower risk of MACE (compared to determining risks with risk scores) at 1 year of admission

CONTACTS AND LOCATIONS:
Overall Officials: Aleem Khand, MbChB,MRCP, Principal Investigator — Aintree University Hospital NHS Trust, Liverpool Heart and Chest Hospital NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
All data anonymised and will be analysed accordingly. Results of the study will be published once analysis completed

REFERENCES:
- [Derived] Khand A, Frost F, Grainger R, Fisher M, Chew P, Mullen L, Patel B, Obeidat M, Albouaini K, Dodd J. Identification of high-risk non-ST elevation myocardial infarction at presentation to emergency department. A prospective observational cohort study in North West England. BMJ Open. 2020 Jun 8;10(6):e030128. doi: 10.1136/bmjopen-2019-030128. PMID 32518208